CLINICAL TRIAL: NCT02421991
Title: Telephone-Delivered Interventions for Smoking Cessation
Acronym: TALK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Consumer Wellness Solutions (Industry); National Institute on Drug Abuse (NIDA) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8298; NCI-2018-02635 (Registry Identifier: NCI / CTRP); RG1001154 (Other: Fred Hutch/University of Washington Cancer Consortium); R01DA038411 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2019-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TALK study group (Experimental): This is the experimental arm of the study. This includes 5 weekly sessions of experimental therapy via telephone. Therapy description withheld to protect the integrity of the study.
  Interventions: Behavioral: Telephone Delivered Intervention
- TALK control group (Active Comparator): This is the control arm of the study. This includes 5 weekly sessions of control therapy via telephone.Therapy description withheld to protect the integrity of the study.
  Interventions: Behavioral: Telephone Delivered Intervention

INTERVENTIONS:
Behavioral: Telephone Delivered Intervention

SUMMARY:
The purpose of this study is to demonstrate that Acceptance and Commitment Therapy's (ACT) implementation outcomes are at least as good as those of traditional cognitive behavioral therapy (CBT).

ELIGIBILITY:
Inclusion Criteria:

1. ages 18 and older
2. smokes at least ten cigarettes per day (to be eligible for NRT) and has done so for at least the past 12 months
3. wants to quit smoking in the next 30 days
4. if concurrently using any other nicotine or tobacco products wants to quit using them within the next 30 days
5. willing to be randomly assigned to either group
6. willing and able to speak and read in English
7. willing and medically eligible to use NRT
8. resides in the U.S., and expects to continue for at least 12 months
9. not participating in other smoking cessation interventions (including our own intervention trials)
10. has regular access to a telephone.

Exclusion Criteria:

The exclusion criteria are opposite of the inclusion criteria listed above.

In addition we will exclude:

1. anyone who is pregnant or breast feeding
2. has had a heart attack in the past 30 days
3. has unstable angina
4. has evidence of arrhythmia in the past 6 months
5. has a history of severe skin reaction to adhesive patches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1275 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
30 day point prevalence abstinence | 12 months
  No smoking in the past 30 days, as reported at 12 month post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Bricker, Ph.D., Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700